CLINICAL TRIAL: NCT02394236
Title: Continuous vs. Interval Exercise Training on Oxygen Uptake Efficiency Slope in Patients With Coronary Artery Disease
Brief Title: Aerobic Exercise and Oxygen Uptake Efficiency Slope in Coronary Artery Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital TotalCor (Other)
Responsible Party: Principal Investigator, Danilo Marcelo Leite do Prado, Danilo ML Prado, Prof.PHD, Hospital TotalCor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 66/2011
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Coronary Artery Disease
Keywords: exercise training
MeSH Terms: conditions — Coronary Artery Disease | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous exercise training (Experimental): The continuous exercise training was performed on a treadmill with a 50-minutes duration and intensity at ventilatory anaerobic threshold.
  Interventions: Other: Aerobic exercise training
- interval exercise training (Experimental): The interval exercise training consisted of 7 sets of 3 minutes at respiratory compensation point and 7 sets of 3 minutes of exercise at moderate intensity corresponding to the ventilatory anaerobic threshold totaling 42 minutes
  Interventions: Other: Aerobic exercise training

INTERVENTIONS:
Other: Aerobic exercise training — The continuous exercise training was performed on a treadmill with a 50-minutes duration and intensity at ventilatory anaerobic threshold.
  The interval exercise training consisted of 7 sets of 3 minutes at respiratory compensation point and 7 sets of 3 minutes of exercise at moderate intensity corresponding to the ventilatory anaerobic threshold totaling 42 minutes
  Other Names: continuos training; interval training

SUMMARY:
Thus, the purpose of the present study was to evaluate the effects of continuos exercise training (CET) and interval exercise trainining (IET) on oxygen uptake efficiency slope (OUES) in patients with coronary artery disease.

DETAILED DESCRIPTION:
The oxygen uptake efficiency slope (OUES) is a submaximal index that incorporates cardiovascular, peripheral and pulmonary factors that determine ventilatory response to exercise. There is scarce information about the effects of the mode and intensity of exercise training on OUES in patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* stable coronary artery disease diagnosed by coronary angiography

Exclusion Criteria:

* unstable angina pectoris,
* complex ventricular arrhythmias,
* pulmonary congestion and
* orthopaedic or neurological limitations to exercise

Ages: 49 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
The oxygen uptake efficiency slope | up to 3 months
  The oxygen uptake efficiency slope (OUES) is a submaximal index that incorporates cardiovascular, peripheral and pulmonary factors that determine ventilatory response to exercise.